CLINICAL TRIAL: NCT07095608
Title: Defining TRPV4 Contribution of Schwann Cells to Oral Cancer Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25-00531; 1K23DE034496-01 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Oral Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Mouth Neoplasms; Carcinoma, Squamous Cell | interventions — Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Cancer Subjects (Experimental): Oral cancer patients will be tested for pressure and stretch sensitivity. Pressure sensitivity will be evaluated with a digital pressure algometer by applying the probe tip to the site of cancer in oral cancer patients.
  Stretch sensitivity will be evaluated with visual analog scale recording of pain scores associated with tongue range of motions in oral cancer patients.
  Interventions: Behavioral: Pressure and stretch sensitivity testing
- Healthy Subjects (Active Comparator): Healthy subjects will be tested for pressure and stretch sensitivity. Pressure sensitivity will be evaluated with a digital pressure algometer by applying the probe tip to the tongues of healthy subjects.
  Stretch sensitivity will be evaluated with visual analog scale recording of pain scores associated with tongue range of motions in healthy subjects.
  Interventions: Behavioral: Pressure and stretch sensitivity testing

INTERVENTIONS:
Behavioral: Pressure and stretch sensitivity testing — We will measure pressure sensitivity by applying gradual pressure (50 kPa/s) at the site of testing using a digital pressure algometer. In healthy subjects, we will perform these measurements on the lateral tongue on the left and the right side. In cancer patients, we will first test on the unaffected contralateral matched site and then at the site of the cancer. We will define pressure sensitivity as the mean of three threshold measurements.
  For measuring stretch sensitivity, we will use a visual analog scale (VAS) recording of pain scores associated with tongue stretching. Participants will be asked to perform tongue range of motions (ROM): protrusion, elevation, right and left lateralization, and rate sensitivity score on the VAS scale after holding the tongue in position for five seconds. We will define stretch sensitivity as the sum of VAS scores for protrusion, elevation, right and left lateralization.

SUMMARY:
This is a prospective study involving human participants. Pressure and stretch sensitivity measures between oral cancer patients and healthy subjects will be compared. Pain stimulation will be conducted on the site of the cancer in 40 oral cancer patients, and on the tongue in 40 healthy volunteers, using pressure and stretch sensitivity tests.

DETAILED DESCRIPTION:
Oral cancer, particularly squamous cell carcinoma (SCC), represents nearly 90% of all head and neck cancers. Most patients with oral cancer experience functional pain caused by pressure at the cancer site, along with discomfort from stretching during activities like talking, drinking, and swallowing. However, the intensity and nature of this pain can vary significantly among individual patients. Currently, there are no effective treatments available to relieve pain associated with oral cancer.

The current hypothesis regarding the cause of oral cancer pain suggests that oral cancers release pain mediators that sensitize and activate receptors on sensory nerves associated with cancer. Mechanosensitive ion channels, such as TRPV4, PIEZO1, and PIEZO2, are activated by pressure and stretch, and have been implicated in pathological pain. Preclinical studies show that mice lacking TRPV4 have impaired pressure sensation, and inhibiting TRPV4 in models of oral cancer reduces mechanical pain. TRPV4 is expressed in various cell types, including epithelial cells, fibroblasts, neurons, and Schwann cells, which are the glial cells that ensheathe the axons of sensory neurons. Cancer cells and Schwann cells interact reciprocally, promoting cancer growth and pain. Preliminary data indicate that Schwann cells isolated from the trigeminal nerve fibers innervating the cancers of oral cancer patients express functional TRPV4. In human Schwann cells, the activation of TRPV4 mediates mechanosensitivity. A TRPV4 inhibitor currently in clinical trials has been well-tolerated by patients and has demonstrated a good safety profile. A better understanding of TRPV4's role in oral cancer pain holds significant promise for the development of TRPV4 antagonists as new analgesics for alleviating pain in oral cancer patients.

There is a lack of published data regarding the effects of pressure and stretch on pain phenotypes in patients with oral cancers. This gap significantly hinders our understanding of the mechanisms underlying oral cancer pain. By quantitatively assessing the pressure and stretch sensitivities experienced by these patients, the investigators can gain valuable insights into the origins of their pain. In this proposal, the investigators hypothesize that the quality of pain experienced by oral cancer patients is influenced by the activation levels of mechanosensitive ion channels at the site of the cancer. The investigators will conduct sensitivity tests for pressure and stretch on oral cancer patients and compare the patients' sensitivities with those of healthy subjects. Furthermore, the investigators will evaluate the correlation between pressure and stretch sensitivity scores in oral cancer patients.

The investigators propose that the degree of pressure and stretch sensitivities experienced by oral cancer patients is quantifiable and depends on the functional expression of TRPV4 on Schwann cells.

ELIGIBILITY:
Inclusion Criteria:

For healthy subjects to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, at least 18 years of age
* In good general health as evidenced by medical history

For oral cancer patients to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, at least 18 years of age
* Biopsy-proven squamous cell carcinoma (SCC) of the oral cavity that requires surgical resection
* Lesion is at least 1 cm in greatest surface dimension

Exclusion Criteria:

* Healthy subjects who meet any of the following criteria will be excluded from participation in this study:

  * Clinically and/or histologically proven oral pre-cancer, oral cancer
  * Pregnancy or lactation (Female subjects of child-bearing potential will have a rapid urine pregnancy test)
  * Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Oral cancer patients who meet any of the following criteria will be excluded from participation in this study:

* History of prior surgical, chemotherapeutic, or radiation treatment for head and neck cancer
* Pregnancy or lactation
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

For participants with impaired kidney function (chronic kidney/renal disease) who wish to participate in the proposed research study, consultation with their primary care provider will be done prior to enrollment to determine safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Pressure sensitivity | Baseline
  Pressure pain thresholds will be measured in kilopascals with a digital pressure algometer. The average of three measurements will be used to determine each threshold. Lower thresholds signify higher pain levels.
Stretch sensitivity | Baseline
  Stretch sensitivity will be evaluated by assessing pain or discomfort associated with tongue range of motions (tongue protrusion, tongue elevation, right lateralization and left lateralization).To measure stretch sensitivity, visual analog scale (VAS) scores for participants' pain associated with tongue stretching will be recorded. Participants will perform tongue range of motions (ROM): protrusion, elevation, and right and left lateralization, and they will rate their sensitivity on the VAS scale after holding each position for five seconds. Subjects will also rate the quality of their pain. Stretch sensitivity will be defined as the sum of VAS scores for protrusion, elevation, and right and left lateralization. The VAS goes from 0-100, 0 representing no pain and 100 representing the most intense pain imaginable.

SECONDARY OUTCOMES:
To determine whether patients with lower pressure pain thresholds report higher pain scores on the visual analog scale after tongue stretching. | Baseline
  Pressure pain thresholds will be measured in kilopascals with a digital pressure algometer. The average of three measurements will be used to determine each threshold. Lower thresholds signify higher pain levels.
  The tongue stretch questionnaire records the total VAS pain scores for lingual range of motion. Higher scores indicate more pain.
  The dependent variables of the pressure and stretch tests will be evaluated for a linear relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Schmidt, DDS, Principal Investigator — NYU College of Dentistry
Locations (1):
- NYU College of Dentistry, New York, New York, United States

REFERENCES:
- [Background] Gormley M, Creaney G, Schache A, Ingarfield K, Conway DI. Reviewing the epidemiology of head and neck cancer: definitions, trends and risk factors. Br Dent J. 2022 Nov;233(9):780-786. doi: 10.1038/s41415-022-5166-x. Epub 2022 Nov 11. PMID 36369568
- [Background] Viet CT, Schmidt BL. Biologic mechanisms of oral cancer pain and implications for clinical therapy. J Dent Res. 2012 May;91(5):447-53. doi: 10.1177/0022034511424156. Epub 2011 Oct 4. PMID 21972258
- [Background] Szczot M, Liljencrantz J, Ghitani N, Barik A, Lam R, Thompson JH, Bharucha-Goebel D, Saade D, Necaise A, Donkervoort S, Foley AR, Gordon T, Case L, Bushnell MC, Bonnemann CG, Chesler AT. PIEZO2 mediates injury-induced tactile pain in mice and humans. Sci Transl Med. 2018 Oct 10;10(462):eaat9892. doi: 10.1126/scitranslmed.aat9892. PMID 30305456
- [Background] Nilius B, Voets T. The puzzle of TRPV4 channelopathies. EMBO Rep. 2013 Feb;14(2):152-63. doi: 10.1038/embor.2012.219. Epub 2013 Jan 11. PMID 23306656
- [Background] Mikesell AR, Isaeva E, Schulte ML, Menzel AD, Sriram A, Prahl MM, Shin SM, Sadler KE, Yu H, Stucky CL. Increased keratinocyte activity and PIEZO1 signaling contribute to paclitaxel-induced mechanical hypersensitivity. Sci Transl Med. 2024 Dec 11;16(777):eadn5629. doi: 10.1126/scitranslmed.adn5629. Epub 2024 Dec 11. PMID 39661703
- [Background] Suzuki M, Mizuno A, Kodaira K, Imai M. Impaired pressure sensation in mice lacking TRPV4. J Biol Chem. 2003 Jun 20;278(25):22664-8. doi: 10.1074/jbc.M302561200. Epub 2003 Apr 13. PMID 12692122
- [Background] Mulpuri Y, Tu NH, Inoue K, Harden G, Nicholson SJ, Seenauth A, Huang Y, Escobar KG, Moayedi Y, Bunnett NW, Albertson DG, Schmidt BL. TRPV4 activation in Schwann cells mediates mechanically induced pain of oral cancer. Front Pain Res (Lausanne). 2025 Mar 12;6:1532885. doi: 10.3389/fpain.2025.1532885. eCollection 2025. PMID 40144515
- [Background] Salvo E, Saraithong P, Curtin JG, Janal MN, Ye Y. Reciprocal interactions between cancer and Schwann cells contribute to oral cancer progression and pain. Heliyon. 2019 Feb 15;5(2):e01223. doi: 10.1016/j.heliyon.2019.e01223. eCollection 2019 Feb. PMID 30815600
- [Background] Goyal N, Skrdla P, Schroyer R, Kumar S, Fernando D, Oughton A, Norton N, Sprecher DL, Cheriyan J. Clinical Pharmacokinetics, Safety, and Tolerability of a Novel, First-in-Class TRPV4 Ion Channel Inhibitor, GSK2798745, in Healthy and Heart Failure Subjects. Am J Cardiovasc Drugs. 2019 Jun;19(3):335-342. doi: 10.1007/s40256-018-00320-6. PMID 30637626